CLINICAL TRIAL: NCT03153436
Title: The Effect of In-vitro Myoinositol Supplementation of Human Sperm on the Outcome of Cryopreservation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Collaborators: Ajyal Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Alaa El-Dein Hasan, M.B.B.Ch., Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SPMYO001
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Myoinositol; Cryopreservation; Human; Sperm
MeSH Terms: interventions — Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal S.A group (Active Comparator): Infertile men with normal semen analysis. each sample is divided into 2 identical aliquots: one aliquot (Myo aliquot) is supplied with myoinositol, The other aliquot is left as it is (control aliquot).
  Interventions: Biological: Myoinositol
- Abnormal S.A group (Active Comparator): Infertile men with abnormal semen analysis. each sample is divided into 2 identical aliquots: one aliquot (Myo aliquot) is supplied with myoinositol, The other aliquot is left as it is (control aliquot).
  Interventions: Biological: Myoinositol

INTERVENTIONS:
Biological: Myoinositol

SUMMARY:
The objective of this study is to evaluate the effect of in-vitro myoinositol supplementation of human sperm on the outcome of cryopreservation.

DETAILED DESCRIPTION:
Sperm cryopreservation is considered the most valuable and used way to preserve male reproductive function. Unfortunately, osmotic effects of freezing and thawing during the cryopreservation process negatively affect sperm morphology and motility .

Myoinositol is the most biologically important form of inositol in nature. In male reproductive system, myoinositol appears to regulate sperm motility, capacitation and acrosomal reaction.

The objective of this study is to evaluate the effect of in-vitro myoinositol supplementation of human sperm on the outcome of cryopreservation.

ELIGIBILITY:
Inclusion Criteria:

* Infertile men with normal or abnormal semen analysis

Exclusion Criteria:

* Azoospermic samples

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Cryo-survival rate | 7 months
  Post-thawing cryo-survival rates of both aliquots ( myo and control) are compared in both groups (A and B).

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, M.D., Study Director — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ackerman DR. The effect of cooling and freezing on the aerobic and anaerobic lactic acid production of human semen. Fertil Steril. 1968 Jan-Feb;19(1):123-8. doi: 10.1016/s0015-0282(16)36552-9. No abstract available. PMID 4952185
- [Background] Anger JT, Gilbert BR, Goldstein M. Cryopreservation of sperm: indications, methods and results. J Urol. 2003 Oct;170(4 Pt 1):1079-84. doi: 10.1097/01.ju.0000084820.98430.b8. PMID 14501696
- [Background] Araki Y, Yao T, Asayama Y, Matsuhisa A, Araki Y. Single human sperm cryopreservation method using hollow-core agarose capsules. Fertil Steril. 2015 Oct;104(4):1004-1009. doi: 10.1016/j.fertnstert.2015.06.043. Epub 2015 Jul 21. PMID 26207962
- [Background] Bahat A, Eisenbach M. Human sperm thermotaxis is mediated by phospholipase C and inositol trisphosphate receptor Ca2+ channel. Biol Reprod. 2010 Mar;82(3):606-16. doi: 10.1095/biolreprod.109.080127. Epub 2009 Dec 2. PMID 19955332
- [Background] Beemster P, Groenen P, Steegers-Theunissen R. Involvement of inositol in reproduction. Nutr Rev. 2002 Mar;60(3):80-7. doi: 10.1301/00296640260042748. PMID 11908744
- [Background] Oberoi B, Kumar S, Talwar P. Study of human sperm motility post cryopreservation. Med J Armed Forces India. 2014 Oct;70(4):349-53. doi: 10.1016/j.mjafi.2014.09.006. Epub 2014 Oct 16. PMID 25382909